CLINICAL TRIAL: NCT07110181
Title: A Randomized Controlled Trial Evaluating the Efficacy of a Blended Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Chinese Adolescents With Non-Suicidal Self-Injury
Brief Title: Blended Unified Protocol for Chinese Adolescents With Non-Suicidal Self-Injury: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Jun Ou (Other)
Responsible Party: Sponsor-Investigator, Jian-Jun Ou, professor, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2024193
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Non-suicidal Self-injury (NSSI)
Keywords: non-suicidal self-injury; adolescent
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UP-A + Treatment as Usual (Experimental): Participants receive standard psychiatric care (e.g., pharmacotherapy) plus a blended version of the Unified Protocol for Adolescents (UP-A), which includes both face-to-face and online sessions over 8 weeks.
  Interventions: Behavioral: a blended version of the Unified Protocol for Adolescents (UP-A); Drug: Standard psychiatric treatment
- Treatment as Usual (Active Comparator): Participants in the control group will receive standard psychiatric care as provided by their treating clinicians, including pharmacotherapy as appropriate. No additional psychological intervention will be provided during the study period.
  Interventions: Drug: Standard psychiatric treatment

INTERVENTIONS:
Behavioral: a blended version of the Unified Protocol for Adolescents (UP-A) — The blended UP-A includes 8 weekly modules, 6 of which (Modules 2 - 7)are online self-guided sessions. The online self-guided sessions will last approximately 45 minutes each. Over the course of these 6 weeks, participants will also have 6 therapist-guided online sessions via videoconference, each lasting 30 minutes. Two face-to-face individual sessions are scheduled, one at the beginning of each (Module 1) and one at the end (Module 8), each with an expected duration of 90 minutes.
  Arms: UP-A + Treatment as Usual
Drug: Standard psychiatric treatment — Participants in the control group will receive treatment as usual, including pharmacotherapy and routine clinical follow-up, as determined by their treating psychiatrists.

SUMMARY:
This study is an open-label, randomized controlled trial evaluating the efficacy of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) in reducing non-suicidal self-injury (NSSI) among Chinese adolescents. This program is an annualized cognitive-behavioral therapy designed for adolescents aged 12-17 years who engage in non-suicidal self-injury behavior. Its primary goal is to reduce the intensity and frequency of distressing emotional experiences by teaching adolescents how to confront and respond to these emotions in more adaptive ways. In turn, this helps reduce self-injury impulses and behaviors. The UP-A is adapted to the Chinese cultural context and delivered as a blended treatment, combining face-to-face and online sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 12 and 17 years;
2. Engaged in non-suicidal self-injury (NSSI) at least 5 times in the past 12 months, with at least 1 episode in the past month;
3. Minimum education level of primary school or above;
4. Participant and guardian fully understand the research content and agree to participate, with signed informed consent provided.

Exclusion Criteria:

1. Suicide attempts in the past month or a score of ≥17 on the MINI National Neuropsychiatric Interview for Children (MINI KID 5.0), indicating a high risk of suicide;
2. Diagnosis of a psychotic disorder, autism spectrum disorder, or other serious neurodevelopmental disorders according to the DSM-5;
3. Presence of severe physical illness or other medical conditions that may affect the completion of treatment and evaluation;
4. Currently receiving other professional psychotherapy or participating in another NSSI intervention study;
5. Received 5 or more sessions of cognitive behavioral therapy (CBT) in the past 5 years;
6. Having received electroconvulsive therapy (ECT) within the past 6 months.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Non-suicidal self-injury behavior | Up to 3 months post-baseline (measured at baseline, 1, 2, and 3 months)
  The Adolescent Self-Harm Behavior Scale includes 18 items describing forms of self-harm. The scale is divided into two dimensions: frequency and severity of self-harm. Self-harm frequency is scored on a 4-point scale (0-3), with the following categories: 0 times, 1 time, 2-4 times, and more than 5 times. The severity of physical injury is scored on a 5-point scale (0-4), with the following categories: none, mild, moderate, severe, and extremely severe. The product of frequency and injury severity for each item is used as the overall score for NSSI, with higher scores indicating more severe NSSI behavior.

SECONDARY OUTCOMES:
Depression | Up to 3 months post-baseline (measured at baseline, 1, 2, and 3 months)
  The Patient Health Questionnaire-9 (PHQ-9) was used to measure depression levels. This nine-item scale rates each item on a four-point scale from 0 ("not at all") to 3 ("nearly every day"), with total scores ranging from 0 to 27. Higher scores indicate greater depression severity.
Anxiety | Up to 3 months post-baseline (measured at baseline, 1, 2, and 3 months)
  The Generalized Anxiety Disorder-7 (GAD-7) was used to assess anxiety levels of participants. This seven-item scale also employs a four-point scoring system from 0 ("not at all") to 3 ("nearly every day"), with higher scores reflecting greater anxiety severity.

OTHER OUTCOMES:
Neuroticism | Up to 3 months post-baseline (measured at baseline, 1, 2, and 3 months)
  The Neuroticism subscale from the Neuroticism-Extraversion-Openness Five-Factor Inventory was selected to measure neuroticism. The Neuroticism subscale consists of 12 items, rated on a 5-point Likert scale. Higher scores indicate a stronger tendency toward neuroticism in the individual.
Emotion regulation strategies | Up to 3 months post-baseline (measured at baseline, 1, 2, and 3 months)
  The Emotion Regulation Questionnaire (ERQ) is used to measure participants' emotional regulation strategies. It consists of 10 items, divided into two dimensions: cognitive reappraisal and expressive suppression. Each item is rated on a 7-point scale, with higher scores indicating a stronger tendency to use the corresponding emotional regulation strategy.
Emotion dysregulation | Up to 3 months post-baseline (measured at baseline, 1, 2, and 3 months)
  Difficulties in Emotion Regulation Scale (DERS) is used to assess the participants' emotional regulation abilities. It consists of 36 items across 6 dimensions, with higher total scores indicating a higher level of emotional dysregulation. The dimensions include: emotional awareness, emotional acceptance, impulse control, emotional understanding, goal-directed behavior, and strategy use.
Distress tolerance | Up to 3 months post-baseline (measured at baseline, 1, 2, and 3 months)
  The Distress Tolerance Scale (DTS) is a 15-item measure of an individual's perceived ability to withstand negative emotions. Items are answered on a five-point Likert scale ranging from 1 = strongly agree to 5 = strongly disagree. Traditionally, high DTS-global distress intolerance scores reflect a heightened ability to tolerate distress, whereas low total scores represent distress intolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No